CLINICAL TRIAL: NCT02324894
Title: Initial Evaluation of Ultra FAST Breast Magnetic Resonance in Breast Cancer Screening: Comparative Study With Mammography and Ultrasound.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was never initiated.
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Dr Divano Luisa, Head of the Radiology Department, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-FastMRI-BCS
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: screening; MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI screening (Other): Diagnostic screening. The normal eligible screening population will first undergo a mammography, then an echography screening followed by a fast MRI screening.
  Interventions: Procedure: MRI screening

INTERVENTIONS:
Procedure: MRI screening — Diagnostic screening. The normal eligible screening population will first undergo a mammography, then an echography screening followed by a fast MRI screening.

SUMMARY:
Mammography remains an imperfect screening test especially in women with extremely dense breast tissue, missing biologically aggressive cancers especially in younger population and picking up indolent cancers that do not need treatment.

The most sensitive test for breast cancer detection at our disposal is magnetic resonance imaging (MRI). The preliminary study of Dr Kuhl provide strong arguments that Ultra FAST Breast Magnetic Resonance is suitable for breast cancer screening with high sensitivity and specificity values.

Data clearly demonstrates that FAST breast MRI could be the standard for breast cancer screening: it is safe, does not induce cancers, and can find more cancers than mammography.

However this study was performed in women with low to moderately increased risk.The value of FAST Breast Magnetic Resonance in normal screening population has to be assessed before a modification of current strategy of breast cancer screening with mammography.

ELIGIBILITY:
Inclusion Criteria:

* Women referred for routine breast cancer screening

Exclusion Criteria:

* Disabled women (eg, unable to stand)
* Pregnant women
* Allergy to Gadolinium

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
ACR five point rating scale for mammography images | 24h
  Two views (craniocaudal and mediolateral oblique) will be obtained of each breast with digital mammography by using a commercially available system. The reader will first interpret the digital mammography using a dedicated workstation.The radiologist will rate the images from each examination by using a standardized ACR five-point rating scale. Furthermore, if a reader records a positive score (>2), mammographic features have to be specified (localization, number of ACR>2 lesions,using predefined evaluation form). Scores are recorded directly into the PACS database and locked after each reading session.
ACR five point rating scale for echography images | 24h
  After the digital mammography, the same reader will perform Ultrasound of both breasts using the transmitter of 10-13 MHertz (Acuson Antares (Siemens)). The reader will then interpret the ultrasound images using the same methodology as for digital mammography, described above (ACR five point rating scale).
ACR five point rating scale for MRI imaging | 24h
  The same day, the Ultra FAST Breast Magnetic Resonance will be performed on 3T unit with 8 channel dedicated breast coil. Sequences: 3 Dimensional Gradient echo with Fat Saturation before and after Gadolinium injection (acquisition time 2 minutes). Initial post processing: MPR and automatic subtraction. The reader has to assess the MRI images using the same methodology as for digital mammography, according to the American College of Radiology Breast Imaging Reporting and Data System.

CONTACTS AND LOCATIONS:
Overall Officials: Tadeusz Stadnik, MD, PhD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Tabar L, Vitak B, Chen TH, Yen AM, Cohen A, Tot T, Chiu SY, Chen SL, Fann JC, Rosell J, Fohlin H, Smith RA, Duffy SW. Swedish two-county trial: impact of mammographic screening on breast cancer mortality during 3 decades. Radiology. 2011 Sep;260(3):658-63. doi: 10.1148/radiol.11110469. Epub 2011 Jun 28. PMID 21712474
- [Background] Kopans DB. Arguments against mammography screening continue to be based on faulty science. Oncologist. 2014 Feb;19(2):107-12. doi: 10.1634/theoncologist.2013-0184. PMID 24536051
- [Background] Miller AB, Wall C, Baines CJ, Sun P, To T, Narod SA. Twenty five year follow-up for breast cancer incidence and mortality of the Canadian National Breast Screening Study: randomised screening trial. BMJ. 2014 Feb 11;348:g366. doi: 10.1136/bmj.g366. PMID 24519768
- [Background] Biller-Andorno N, Juni P. Abolishing mammography screening programs? A view from the Swiss Medical Board. N Engl J Med. 2014 May 22;370(21):1965-7. doi: 10.1056/NEJMp1401875. Epub 2014 Apr 16. No abstract available. PMID 24738641
- [Background] Morris EA. Diagnostic breast MR imaging: current status and future directions. Magn Reson Imaging Clin N Am. 2010 Feb;18(1):57-74. doi: 10.1016/j.mric.2009.09.005. PMID 19962093
- [Background] Kuhl CK, Schrading S, Strobel K, Schild HH, Hilgers RD, Bieling HB. Abbreviated breast magnetic resonance imaging (MRI): first postcontrast subtracted images and maximum-intensity projection-a novel approach to breast cancer screening with MRI. J Clin Oncol. 2014 Aug 1;32(22):2304-10. doi: 10.1200/JCO.2013.52.5386. Epub 2014 Jun 23. PMID 24958821
- [Background] Berg WA, Zhang Z, Lehrer D, Jong RA, Pisano ED, Barr RG, Bohm-Velez M, Mahoney MC, Evans WP 3rd, Larsen LH, Morton MJ, Mendelson EB, Farria DM, Cormack JB, Marques HS, Adams A, Yeh NM, Gabrielli G; ACRIN 6666 Investigators. Detection of breast cancer with addition of annual screening ultrasound or a single screening MRI to mammography in women with elevated breast cancer risk. JAMA. 2012 Apr 4;307(13):1394-404. doi: 10.1001/jama.2012.388. PMID 22474203
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB, Lehrer D, Bohm-Velez M, Pisano ED, Jong RA, Evans WP, Morton MJ, Mahoney MC, Larsen LH, Barr RG, Farria DM, Marques HS, Boparai K; ACRIN 6666 Investigators. Combined screening with ultrasound and mammography vs mammography alone in women at elevated risk of breast cancer. JAMA. 2008 May 14;299(18):2151-63. doi: 10.1001/jama.299.18.2151. PMID 18477782
- [Background] Kuhl C, Weigel S, Schrading S, Arand B, Bieling H, Konig R, Tombach B, Leutner C, Rieber-Brambs A, Nordhoff D, Heindel W, Reiser M, Schild HH. Prospective multicenter cohort study to refine management recommendations for women at elevated familial risk of breast cancer: the EVA trial. J Clin Oncol. 2010 Mar 20;28(9):1450-7. doi: 10.1200/JCO.2009.23.0839. Epub 2010 Feb 22. PMID 20177029
- [Background] Kuhl CK. Why do purely intraductal cancers enhance on breast MR images? Radiology. 2009 Nov;253(2):281-3. doi: 10.1148/radiol.2532091401. No abstract available. PMID 19864520
- [Background] Feig S. Cost-effectiveness of mammography, MRI, and ultrasonography for breast cancer screening. Radiol Clin North Am. 2010 Sep;48(5):879-91. doi: 10.1016/j.rcl.2010.06.002. PMID 20868891